CLINICAL TRIAL: NCT00982904
Title: Randomized, Double-blind, Placebo-controlled Study of the Tolerability, and Pharmacokinetics of Fexinidazole After Single and Repeated Oral Ascending Doses, Completed by a Comparative Bioavailability Study of an Oral Suspension Versus a Tablet and an Exploratory Assessment of Food Effect, in Healthy Male Volunteers
Brief Title: Human African Trypanosomiasis: First in Man Clinical Trial of a New Medicinal Product, the Fexinidazole
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DNDiFEX001
Record Dates: First submitted 2009-09-22; First posted 2009-09-23 (Estimated); Last update posted 2017-04-06 (Actual); Status verified 2017-04

CONDITIONS: Human African Trypanosomiasis
Keywords: neglected disease; africa; new drug; oral drug; parasite
MeSH Terms: conditions — Neglected Diseases | interventions — fexinidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fexinidazole (Experimental)
  Interventions: Drug: Fexinidazole/Placebo
- Placebo (Placebo Comparator)
  Interventions: Drug: Fexinidazole/Placebo

INTERVENTIONS:
Drug: Fexinidazole/Placebo

SUMMARY:
This study is aimed at assessing the tolerability and pharmacokinetic parameters of the fexinidazole in healthy volunteers. In animal models of both acute and chronic experimental Trypanosomiasis infections, fexinidazole shows highly promising efficacy.

DETAILED DESCRIPTION:
The present study is designed to obtain safety, tolerability and PK data after single and multiple oral administration of increasing doses of fexinidazole in healthy male sub-Saharan African subjects. This study will also assess the relative bioavailability of fexinidazole administered as a tablet in comparison with oral suspension, and to assess the impact of concomitant food intake on the relative bioavailability of fexinidazole after single oral dose administration.

The study will be divided in 3 successive parts. Study Part I will be a randomized, double-blind, placebo-controlled, single ascending dose study with fexinidazole administered as an oral suspension.

Study Part II will be a comparative bioavailability study of a fexinidazole tablet vs. the oral suspension and assessment of food effect, according to a three-way cross-over design. Clinical part will be conducted in open conditions and bioanalysis in blind conditions.

Study Part III will be a randomized, double-blind, placebo-controlled, multiple ascending dose study with fexinidazole administered either as an oral suspension or as a tablet, depending on Part II results. Dosage regimen will be either q.d. or b.i.d., depending on Part I and Part II results for the unchanged drug and the metabolites. Treatment duration will be 14 days.

Bioanalysis will be performed in open conditions for Study Part I and Study Part III.

ELIGIBILITY:
Inclusion Criteria:

* All subjects to be of sub-Saharan African origins with both parents of sub-Saharan African origins too,
* Male subjects with a body mass index (BMI) calculated as weight in kg/(height in m2) from 18 to 28 kg/m2 at screening,
* Able to communicate well with the Investigator and research staff and to comply with the requirements of the entire study,
* Provision of written informed consent to participate as shown by a signature on the volunteer consent form,
* Light smokers (less than 5 cigarettes per day) or subjects who are non-smokers.
* Normal arterial blood pressure (BP) and pulse rate or, if abnormal, considered not clinically significant by the principal Investigator.
* Registered with the French Social Security in agreement with the French law on biomedical experimentation.

Exclusion Criteria:

* Who on direct questioning and physical examination have evidence of any clinically significant acute or chronic disease, including known or suspected HIV, HBV or HCV infection,
* Who previously received fexinidazole,
* With any clinically significant abnormality following review of pre-study laboratory tests(ASAT, ALAT and ALP must be within normal ranges), vital signs, full physical examination and ECG,
* Who are within the exclusion period defined in the National Register for Healthy Volunteers of the French Ministry of Health,
* Who forfeit their freedom by administrative or legal award or who were under guardianship,
* Unwilling to give their informed consent,
* Who have a positive laboratory test for Hepatitis B surface antigen (HbsAg), or anti-HIV 1/2 or anti- HCV antibodies
* Who have a history of allergy, intolerance or photosensitivity to any drug,
* Who have a history of serious allergy, asthma, allergic skin rash or sensitivity to any drug,
* Who are known or suspected alcohol or drug abusers (more than 14 units of alcohol per week, one unit = 8 g or about 10 mL of pure alcohol),
* Who drink more than 8 cups daily of beverage containing caffeine,
* Who have a positive laboratory test for urine drug screening
* Who have undergone surgery or have donated blood within 12 weeks prior to the start of the study,
* Who have taken any prescribed or over the counter drug (including antacid drug), with the exception of paracetamol (up to 3 g per day) within 2 weeks prior to the first dose administration,
* Who have any clinical condition or prior therapy which, in the opinion of the Investigator, made the subject unsuitable for the study,
* Who participated to any clinical trial with an investigational drug in the past 3 months preceding study entry.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 108 (Actual)
Dates: Start 2009-09; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Occurence of adverse events (AEs) | 8 to 37 days, depending on the part of the study

SECONDARY OUTCOMES:
Pharmacokinetic : measure of blood and urine concentration of fexinidazole, fexinidazole sulfoxide and fexinidazole sulfone in order to determine AUC0-t and Cmax values, for all dose levels | pre-dose, and 0.5, 1, 2, 3, 4, 6, 9, 12, 16, 24, 48, 72, 96, 120, 144 and 168 h post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Lionel Hovsepian, MD, Principal Investigator — SGS Aster; Nathalie Strub-Wourgaft, MD, Study Chair — Drugs for Neglected Diseases initiative
Locations (1):
- SGS Aster, Paris, France

REFERENCES:
- See also: Sponsor Website — http://www.dndi.org
- See also: Publication combining NCT01340157 & NCT01483170 — http://www.dndi.org/wp-content/uploads/2009/06/ClinicalPK_Tarral_FexinidazoleHAT_2014.pdf
- Available data/document: Publication of results — http://www.dndi.org/wp-content/uploads/2009/06/ClinicalPK_Tarral_FexinidazoleHAT_2014.pdf — Publication of results